CLINICAL TRIAL: NCT05130580
Title: Evaluation of a Patient-Specific Decision Aid System for Shared Decision-Making About Breast Reconstruction
Brief Title: Patient-Specific Decision Aid System for Shared Decision Making About Breast Reconstruction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-1176; NCI-2020-11520 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1176 (Other: M D Anderson Cancer Center); R01CA203984 (NIH)
Record Dates: First submitted 2021-09-09; First posted 2021-11-23 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Referral and Consultation; Congresses as Topic; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (educational materials, enhanced consult, decision aid) (Experimental): Patients receive newly-developed educational materials about breast reconstruction and attend an enhanced consultation visit with their plastic surgeon to discuss options for breast reconstruction surgery, during which a decision aid application containing a customized presentation of possible breast reconstruction outcomes is presented. At the end of the consultation visit, patients complete questionnaires about decision-making and psychological well-being. Within 4-6 weeks and 3-6 months after beginning the reconstruction process, patients also complete questionnaires about satisfaction with their breasts, body image, and psychological well-being, and undergo two-dimensional (2D) and 3D imaging of the torso.
  Interventions: Other: Enhanced Consultation; Procedure: Conventional Imaging; Other: Educational Intervention; Other: Questionnaire Administration
- Arm II (educational materials, standard of care consultation) (Active Comparator): Patients receive newly-developed educational materials about breast reconstruction and attend a standard of care consultation visit with their plastic surgeon to discuss options for breast reconstruction surgery. At the end of the consultation visit, patients complete questionnaires about decision-making and psychological well-being. Within 4-6 weeks and 3-6 months after beginning the reconstruction process, patients also complete questionnaires about satisfaction with their breasts, body image, and psychological well-being, and undergo 2D and 3D imaging of the torso.
  Interventions: Other: Standard of Care Consultation; Procedure: Conventional Imaging; Other: Educational Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Enhanced Consultation — Attend an enhanced consultation with decision aid
  Other Names: Consult
  Arms: Arm I (educational materials, enhanced consult, decision aid)
Other: Standard of Care Consultation — Attend standard of care consultation
  Other Names: Consultation
  Arms: Arm II (educational materials, standard of care consultation)
Procedure: Conventional Imaging — Undergo 2D and 3D torso imaging
  Other Names: Conventional CT; Conventional MRI; Conventional US
Other: Educational Intervention — Receive educational materials
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates whether a decision aid application (app) is effective in helping breast reconstruction surgery patients make informed decisions about breast reconstruction surgery. Researchers have created a computer app for breast reconstruction surgery patients that presents images of breast reconstruction outcomes that are customized to the individual patient's treatment options and personal preferences. This decision aid app may help educate patients about how they might look after surgery and answer their questions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate a newly-developed computer application designed to facilitate shared decision making about breast reconstruction for practicability and usability.

SECONDARY OBJECTIVES:

I. To evaluate the effect of the decision aid application measured as the patient's decisional conflict, decision regret, and psychosocial well-being.

II. To evaluate the accuracy of predicted breast reconstruction outcomes to enhance the mathematical and physics-based algorithms for future use.

EXPLORATORY OBJECTIVE:

I. To evaluate patients' aesthetic measures, such as symmetry, breast volume, breast contour and ptosis 3 months after surgery.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive newly-developed educational materials about breast reconstruction and attend an enhanced consultation visit with their plastic surgeon to discuss options for breast reconstruction surgery, during which a decision aid application containing a customized presentation of possible breast reconstruction outcomes is presented. At the end of the consultation visit, patients complete questionnaires about decision-making and psychological well-being. Within 4-6 weeks and 3-6 months after beginning the reconstruction process, patients also complete questionnaires about satisfaction with their breasts, body image, and psychological well-being, and undergo two-dimensional (2D) and 3D imaging of the torso.

ARM II: Patients receive newly-developed educational materials about breast reconstruction and attend a standard of care consultation visit with their plastic surgeon to discuss options for breast reconstruction surgery. At the end of the consultation visit, patients complete questionnaires about decision-making and psychological well-being. Within 4-6 weeks and 3-6 months after beginning the reconstruction process, patients also complete questionnaires about satisfaction with their breasts, body image, and psychological well-being, and undergo 2D and 3D imaging of the torso.

ELIGIBILITY:
Inclusion Criteria:

* MD Anderson patients, age 21 or older
* Planning to undergo either a unilateral or bilateral total, skin-sparing or nipple-sparing mastectomy; or, planning to undergo a unilateral or bilateral modified radical mastectomy
* Considering immediate breast reconstruction at MD Anderson
* Likely to be a suitable candidate for implant-based reconstruction and/or abdominal-tissue based reconstruction as determined by an MD Anderson Plastic Surgery faculty member
* Ambulatory and able to stand unassisted for two minutes (3D imaging system requirement)
* Ability to understand and read English without a translator

Exclusion Criteria:

* Has had a prior consultation with a plastic surgeon to discuss breast reconstruction
* History of breast surgery (i.e., breast reduction, mastopexy, segmental mastectomy, augmentation, reconstruction, but not including biopsy)
* Planning to have a delayed breast reconstruction
* Adjuvant radiation of the breast is indicated at the time of enrollment
* Diagnosis consistent with psychosis (such as schizophrenia, schizoaffective disorder, major depressive disorder [MDD] with psychotic features or steroid induced psychosis) in the chart
* Diagnosis consistent with cognitive impairment such as dementia, cognitive changes with stroke or radiation therapy in the chart
* Documented personality disorder
* Presence of non-medical tattoo on the breast

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Length of consultation visit | up to 90 minutes
Participant's decisional conflict score-Questionnaires | at 6 months post-operation
  Decisional conflict is measured using the Decisional Conflict Scale (DCS). Scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Reece, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center — http://www.mdanderson.org